CLINICAL TRIAL: NCT06389422
Title: Phase II Study of Moderate-dose Hypofractionated Radiotherapy Combined With Pembrolizumab for Hepatocellular Carcinoma With Diffuse Tumor Thrombosis Involved Both Left and Right Liver
Brief Title: Phase II Study of Moderate-dose Hypofractionated RT Combined With Pembrolizumab for HCC With Diffuse Tumor Thrombosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, BO CHEN, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4620
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma; Radiotherapy; Pembrolizumab; Tumor Thrombosis
Keywords: Hepatocellular Carcinoma; Radiotherapy; Pembrolizumab; Tumor Thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Radiotherapy and Pembrolizumab (Experimental): Moderate-dose hypofractionated intensity-modulated radiotherapy with a gross tumor dose of 25Gy/5f and a maximum dose of 35Gy/5f at the tumor center concurrent with Pembrolizumab, followed Pembrolizumab±lenvatinib for maintenance.
  Interventions: Radiation: Moderate-dose Hypofractionated Intensity-modulated Radiotherapy; Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Moderate-dose Hypofractionated Intensity-modulated Radiotherapy — All lesions receive moderate-dose hypofractionated intensity-modulated radiotherapy, with a gross tumor dose of 25Gy/5f, and a maximum dose of 35Gy/5f at the tumor center.
Drug: Pembrolizumab — One week before or during the radiotherapy, patients receive concurrent Pembrolizumab at a dose of 200mg. Subsequently, Pembrolizumab is administered intravenously every 3 weeks. Follow-up examinations are conducted 1-3 months post-radiotherapy. Lenvatinib 4mg may be used for maintenance therapy with Pembrolizumab if there are no contraindications. Maintenance therapy is continued until disease progression or intolerance.

SUMMARY:
This is a single-center, single-arm, open-label study that includes patients meeting the inclusion criteria (liver-GTV volume < 700ml or estimated liver-GTV V5 < 300ml) with hepatocellular carcinoma with diffuse tumor thrombosis involving both left and right lobes. All lesions receive moderate-dose hypofractionated intensity-modulated radiotherapy, with a gross tumor dose of 25Gy/5f, and a maximum dose of 35Gy/5f at the tumor center. One week before or during the radiotherapy, patients receive concurrent Pembrolizumab at a dose of 200mg. Subsequently, Pembrolizumab is administered intravenously every 3 weeks. Follow-up examinations are conducted 1-3 months post-radiotherapy. Lenvatinib 4mg may be used for maintenance therapy with Pembrolizumab if there are no contraindications. Maintenance therapy is continued until disease progression or intolerance. The primary endpoint is median overall survival (mOS), and secondary endpoints include objective response rate (ORR), progression-free survival (PFS), and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed clinically or histopathologically as hepatocellular carcinoma, concurrently with portal vein thrombosis or hepatic vein thrombosis;
2. Age 18-90 years;
3. Liver-GTV volume<700ml or the estimated volume of Liver-GTV receiving less than 5 Gy of irradiation<300ml but the average dose of Liver-GTV needs to be <18Gy;
4. Allowed previous treatment including TACE, RFA, surgery, chemotherapy, targeted therapy, etc., but not including ICIs such as anti-PD-1, anti-PD-L1, or anti-PD-L2 therapies;
5. ECOG performance status 0-2, expected survival greater than 1 month;
6. Allowing patients with distant metastases;
7. Child-Pugh A5, A6, B7 and B8;
8. ALT within 2.5 times the normal upper limit; AST within 2.5 times the normal upper limit; TBIL <60umol/L.
9. No significant abnormalities in the electrocardiogram, no apparent heart failure, and no contraindications for anti-PD-1 treatment;
10. CRE, BUN within 2.5 times the normal upper limit;
11. Hb ≥ 50g/L, ANC ≥ 0.5 × 10^9 /L, PLT ≥ 30 × 10^9 /L; patients with a history of gastrointestinal bleeding must be controlled for more than 2 weeks before enrollment with Hb ≥ 60g/L and a significant rising trend;
12. Patients voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Currently participating in other clinical trials;
2. Previously received abdominal radiotherapy or liver transplantation;
3. Individuals with severe chronic disease conditions affecting vital organs such as the heart, kidneys, or liver;
4. Severe ascites with noticeable symptoms, anticipated to be unrelieved after treatment.
5. Suspected or confirmed drug addiction, medicine abuse,or alcoholism
6. Pregnant or lactating women;
7. Severe mental or neurological disorders
8. Presence of other life-threatening malignancy within the last 3 years before the start of the study (excluding superficial skin cancer, localized low-grade malignant tumor and in situ carcinoma).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Median Overall Survival | 24 months
  Median Overall Survival (mOS) is defined as the median of Overall Survival (OS). OS is defined as the time from the end of radiotherapy to death from any cause

SECONDARY OUTCOMES:
Objective Response Rate | Assessment in 1 to 3 months after radiotherapy
  Treatment response was defined as the best response in 3 months after radiotherapy. ORR is defined as the percentage of patients who met the complete response (CR) or partial response (PR) criteria as defined by the modified Response Evaluation Criteria in Solid Tumors (mRECIST) and RECIST 1.1
Progression-free Survival | 24 months
  Progression-free Survival (PFS) is defined as the time from the end of RT until tumor progression or death from any cause.
Toxicity | up to 24 months
  Toxicity is assessed and graded according to the Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0).
  Toxicity is assessed and graded according to the Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0).
  Toxicity is assessed and graded according to the Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0).
  Toxicity is assessed and graded according to the Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciecnces and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No